CLINICAL TRIAL: NCT05550311
Title: The Investigation of the Effects of Robot-Assisted Rehabilitation on Respiratory Parameters, Dyspnea and Functional Capacity in Individuals With Stroke
Brief Title: Robot-Assisted Rehabilitation in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc.Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 65-22-10
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: robot-assisted training; respiratory parameters
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot group (Experimental): In addition to conventional treatment, an upper extremity robot-assisted rehabilitation program will be applied for 45 minutes a day, two days a week.
  Interventions: Other: Robot-assisted rehabilitation; Other: Conventional rehabilitation
- Control Group (Active Comparator): Participants in this group will be included in a conventional rehabilitation program
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Robot-assisted rehabilitation — In addition to conventional treatment, an upper extremity robot-assisted rehabilitation program. Range of motion exercises will display on the monitor as a game form. There are 4 games available on the computer (airplane game, rabbit shooting game, ball game, and shopping game) and these games can provide exercises for three joints (shoulder, elbow wrist). There are also 3 different levels of resistance apparatus for each joint. People with a full range of motion can do these exercises with resistance. Before starting the rehabilitation, which joint and which movement to do is determined. To the person; After explaining the desired movement and how to play the game shown on the monitor, the exercises are started. The exercises last 45 minutes, during which exercises are performed for the shoulder, elbow, and wrist.
  Arms: Robot group
Other: Conventional rehabilitation — The conventional Rehabilitation Program consists of; range of motion exercises, strengthening exercises, stretching exercises, balance, and walking exercises and Bobath based neurophysiological approaches.

SUMMARY:
Stroke has a high rate of morbidity and mortality worldwide. This disease is the third leading cause of death after ischemic heart disease and cancer. Stroke is also the leading cause of disability in adults. It is known that stroke individuals have not only limb restriction, but also respiratory capacity and exercise capacity. It has been shown in the literature that upper extremity functions are directly related to respiratory capacity. Although it is known that upper extremity training has positive effects on respiratory capacity in stroke individuals, more studies are needed to examine the effects of upper extremity robot-assisted rehabilitation on respiratory capacity. The aim of this study is to examine the effects of upper extremity robot-assisted rehabilitation applied in addition to conventional treatment on respiratory parameters, dyspnea, and functional capacity.

DETAILED DESCRIPTION:
One of the most common complications in stroke patients is pulmonary aspiration and pneumonia, which are associated with respiratory functions being affected. Fluoroscopic examinations of stroke patients showed decreased movement in the diaphragm as well as in other muscles on the affected side. The combination of a decrease in respiratory parameters, weakness in respiratory muscles, and a decrease in diaphragmatic activity can cause dyspnea in individuals even that require minimal effort. The low level of physical activity is accompanied by a decrease in respiratory functions, and the participation of individuals in society decreases. The purpose of stroke rehabilitation is to reduce the complications caused by stroke and to increase the individual's psychological, social, physical, and professional level of independence and functionality to the highest level. Nowadays, stroke rehabilitation can be shaped by a variety of methods. In clinics, robotic rehabilitation is commonly used for stroke patients with the development of the technology. In the literature, studies show the effect of robotic rehabilitation on respiratory parameters, also robot-assisted walking training provides significant improvement in some respiratory parameters and increases aerobic capacity. The aim of this study is to evaluate the effects of upper extremity robot-assisted rehabilitation applied in addition to conventional treatment on respiratory parameters, dyspnea, and functional capacity in individuals with stroke.

ELIGIBILITY:
Inclusion Criteria :

* Between the ages of 18-65,
* Diagnosed with hemorrhagic or ischemic stroke,
* Having a stroke history of at least 3 months,
* Being 16 and above according to the Mini-Mental State Test,
* Three and above according to the Brunnstrom stage,
* Individuals not included in another rehabilitation program will be included.

Exclusion Criteria:

* Chronic cardiac or pulmonary diseases such as COPD, asthma, interstitial lung disease, and heart failure,
* Using tobacco and tobacco products,
* Severe spasticity to prevent robotic rehabilitation (on Modified Ashworth Scale,
* With skin ulcers,
* Non-union or unstable fracture status,
* Individuals with pressure sores will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume 1. second (FEV1)/ Forced vital capacity (FVC) ratio | Change from Baseline Forced expiratory volume 1. second (FEV1)/ Forced vital capacity (FVC) ratio at 6 weeks
  Spirometric evaluation will be performed to determine the FEV1/FVC value of the participants.
Maximal inspiratory pressure | Change from Baseline Maximal inspiratory pressure at 6 weeks
  Mouth pressure will be assessed to document inspiratory muscle strength
Maximal expiratory pressure | Change from Baseline Maximal expiratory pressure at 6 weeks
  Mouth pressure will be assessed to document expiratory muscle strength
Peak Expiratory Flow Rate | Change from Baseline Peak Expiratory Flow Rate at 6 weeks
  Spirometric assessment will be performed to determine participants' peak expiratory flow rate.

SECONDARY OUTCOMES:
Peak cough flow | Change from Baseline Peak cough flow at 6 weeks
  Peak cough flow will be measured in triplicate during the "maximal coughing manoeuvre" with a digital PEFmeter.
6 Minutes Walking Test | Change from Baseline 6 Minutes Walking Test at 6 weeks
  The 6 minutes walk test is a sub-maximal exercises test use to assess aerobic capacity and endurance.
Time Up and Go Test | Change from Baseline Time Up and Go Test at 6 weeks
  The test evaluates the dynamic balance and mobility.
Dyspnea-12 Scale | Change from Baseline Dyspnea-12 Scale at 6 weeks
  The dyspnea perception will be measured with this scale. There are 12 descriptor items on this scale ranging none (0), mild (1), moderate (2) or severe (3). It provides an overall score for breahtlessness severity that incorporates seven physical items and five affective items.
Satisfaction survey | At 6 weeks
  This text is used to assess patients' satisfaction. Evaluation will be scored between c0-5 as a verbal response. 0 = not at all satisfied, 5 = very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, Assoc.Prof., Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared during the publication process if the journal will ask.

REFERENCES:
- [Derived] Okumus B, Akinci B, Aytutuldu GK, Baran MS. Impact of upper extremity robotic rehabilitation on respiratory parameters, functional capacity and dyspnea in patients with stroke: a randomized controlled study. Neurol Sci. 2025 Mar;46(3):1257-1266. doi: 10.1007/s10072-024-07868-z. Epub 2024 Nov 11. PMID 39527236